CLINICAL TRIAL: NCT02974881
Title: HighLife™ Transcatheter Mitral Valve Replacement System for Severe Mitral Regurgitation in Patients at High Surgical Risk
Brief Title: HighLife™ Transcatheter Mitral Valve Replacement System Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HighLife SAS (Industry)
Collaborators: MedPass International (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-2016-01
Record Dates: First submitted 2016-11-11; First posted 2016-11-29 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Mitral Valve Regurgitation; Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transcatheter mitral valve replacement (Experimental): HighLife TMVR System is a novel and innovative approach developed as an alternative treatment for severe MR when medical treatment is maximal and surgical interventions not possible or at high risk. The HighLife TMVR system is composed of a Transcatheter Mitral Valve (TMV), a sub-annular implant (SAI), and their delivery systems and loading tools. The HighLife Valve is a 31 mm mitral bioprosthesis made of a self-expanding Nitinol frame covered with polyester graft and supporting bovine pericardium leaflets. The bioprosthesis is used in conjunction with the Sub-Annular Implant (SAI).
  Interventions: Device: Transcatheter Mitral Valve Replacement

INTERVENTIONS:
Device: Transcatheter Mitral Valve Replacement — Minimally invasive transcatheter mitral valve implantation using the HighLife™ TMVR system

SUMMARY:
Multicenter feasibility study of the HighLife™ TMVR system.

DETAILED DESCRIPTION:
This is an exploratory clinical study designed to evaluate the feasibility, safety and performance of the Highlife TMVR System in a population of patients with severe symptomatic mitral regurgitation, who are not suitable for surgical or approved percutaneous treatments according to the judgement of the Heart Team. The data gathered in this study will allow to evaluate the feasibility of mitral replacement using the HighLife™ TMVR system and characterize the safety and performance profile of the HighLife™ TMVR System.

All patients will be followed periodically up to 12 months after the intervention and long term safety and performance will be collected annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe mitral regurgitation
* New York Heart Association (NYHA) Functional Class II, III or ambulatory IV.
* Patient is under maximally tolerated GDMT (incl. CRT) for at least 3 months
* Multidisciplinary Heart Team consensus that the patient is inoperable or at high-risk for surgical repair/replacement due to significant co-morbid conditions
* Multidisciplinary Heart Team consensus that the patient is not a suitable candidate for other approved percutaneous repair therapy due to anatomical or medical conditions
* Patient meets the anatomical criteria for HighLife valve sizing as determined by CT and TEE

Main Exclusion Criteria:

* Mitral stenosis
* Rheumatic valve disease
* Severe calcifications of the mitral annulus and/or mitral leaflets
* Prior surgical or interventional treatment of the mitral valve
* Unsuitable anatomy for the transapical access
* Unsuitable anatomy of the aorta and ilio-femoral vessels for the transfemoral access
* Untreated clinically significant coronary artery disease requiring revascularization
* LVEF < 30%
* LVEDD > 70mm
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Hypertrophic Obstructive Cardiomyopathy (HOCM)
* Any surgical or interventional procedure (including PCI) done in the past 30 days prior to procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Freedom of major adverse events | at 30 days post procedure
  including:
  * All-cause mortality
  * Myocardial infarction or coronary ischemia requiring PCI or CABG
  * Major stroke
  * Life-threatening bleeding (MVARC scale)
  * Major access and vascular complications
  * Stage 2 or 3 acute kidney injury (includes dialysis)
  * Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
  * Severe hypotension, heart failure or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for ≥ 48H
Continued intended performance of the HighLife™ bioprosthesis | at 30 days post procedure
  defined as the reduction of mitral regurgitation (MR) to either optimal (0+ to trace) or acceptable (reduced by at least 1 grade from baseline with no more than 2+ MR) without significant mitral stenosis (post-procedure EOA ≥ 1.5 cm2 with a transmitral gradient < 5mmHg) and with no greater than mild (1+) paravalvular MR (and without associated hemolysis)
Technical success | immediately after procedure
  defined as alive patient at exit from procedure room, with all of the following:
  * Successful access, delivery and retrieval of the HighLife delivery systems
  * Deployment and correct positioning of the HighLife bioprosthesis
  * Freedom of additional emergency surgery or re-intervention related to the device or access procedure

SECONDARY OUTCOMES:
Device Success (per MVARC definitions) | At 30 days, 6 months and 12 months post procedure
  per MVARC definition
Procedure Success | At 30 days, 6 months and 12 months post procedure
  per MVARC definition
Patient Success | At 30 days, 6 months and 12 months post procedure
  per MVARC definition
Hemodynamic Performance vs. Baseline | At 7 days, 30 days, at 6 months and 12 months and at 2, 3, 4 and 5 years
  Echocardiographic evaluation
Functional Improvement vs. Baseline | At 30 days, 6 months and 12 months
  New York Heart Association Class 6-Minute Walk Test
Quality of Life Improvement vs. Baseline | At 6 months and 12 months
  Kansas City Cardiomyopathy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Collet, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpétrière Institut de Cardiologie
Locations (10):
- France (6):
  - CHRU Lille, Lille
  - Hôpital Privé Jacques Cartier, Massy
  - CHU Nantes, Nantes
  - Groupe Hospitalier Pitié-Salpétrière Institut de Cardiologie, Paris
  - CHU Rennes Pontchaillou, Rennes
  - CHU Toulouse Rangueil, Toulouse
- Germany (4):
  - Universitätsklinikum, Bonn
  - Universitäres Herzzentrum Hamburg GmbH (UHZ), Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum München des Freistaates Bayern, Munich

REFERENCES:
- [Background] Lange R, Piazza N. HighLife transcatheter mitral valve replacement. EuroIntervention. 2016 Sep 18;12(Y):Y81-3. doi: 10.4244/EIJV12SYA22. No abstract available. PMID 27640044
- [Background] Stone GW, Adams DH, Abraham WT, Kappetein AP, Genereux P, Vranckx P, Mehran R, Kuck KH, Leon MB, Piazza N, Head SJ, Filippatos G, Vahanian AS; Mitral Valve Academic Research Consortium (MVARC). Clinical Trial Design Principles and Endpoint Definitions for Transcatheter Mitral Valve Repair and Replacement: Part 2: Endpoint Definitions: A Consensus Document From the Mitral Valve Academic Research Consortium. J Am Coll Cardiol. 2015 Jul 21;66(3):308-321. doi: 10.1016/j.jacc.2015.05.049. PMID 26184623
- [Background] Barbanti M, Piazza N, Mangiafico S, Buithieu J, Bleiziffer S, Ronsivalle G, Scandura S, Giuffrida A, Popolo Rubbio A, Mazzamuto M, Sgroi C, Lange R, Tamburino C. Transcatheter Mitral Valve Implantation Using the HighLife System. JACC Cardiovasc Interv. 2017 Aug 28;10(16):1662-1670. doi: 10.1016/j.jcin.2017.06.046. PMID 28838477